CLINICAL TRIAL: NCT01002521
Title: Molecular and Genetic Analysis of Disturbed Wound Healing in Barbadians With Diabetic Foot Ulcers
Brief Title: Wound Healing In Diabetes (WHy) Study
Acronym: WHy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: The University of The West Indies (Other)
Collaborators: Chronic Disease Research Centre (Unknown); Barbados Diabetes Foundation (Other)
Responsible Party: R.Clive Landis/Principal Investigator, Chronic Disease Research Centre
Other Study IDs: CDRC-WHy-1
Record Dates: First submitted 2009-10-23; First posted 2009-10-27 (Estimated); Last update posted 2009-10-27 (Estimated); Status verified 2009-10

CONDITIONS: Impaired Wound Healing; Diabetes Mellitus
Keywords: Diabetes; vascular; haptoglobin; tumor; necrosis; factor; alpha; traps; impaired; wound; healing; Impaired wound healing in patients with diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus; Neoplasms; Necrosis; Periodic fever, familial, autosomal dominant; Wounds and Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood,Serum,DNA,Urine
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Cases: Persons With Diabetes (PWD) who have current non-healing ulcer(s)
- Controls: Persons With Diabetes (PWD) with no current ulcers and no history of ulcers

SUMMARY:
This observational study aims to identify risk factors and molecular mechanisms of impaired wound healing, to guide better foot care in the diabetic population.

DETAILED DESCRIPTION:
Diabetes is linked with vascular complications of the eye, kidney and foot. Barbadians suffer from an unusually high prevalence of diabetic foot complications, which can cause difficult-to-heal foot ulcers and even lead to amputations of the toes or feet.Studies from the CDRC have indicated alarmingly high rates of amputation and mortality due to diabetic foot in Barbados. The goal of this study is to improve early detection of persons at risk of the vascular complications of diabetes through non-invasive scanning and genetic susceptibility tests.

The general hypothesis to be tested in this study is that persons with diabetes (PWD) and non-healing foot ulcers are more likely to have a disturbed mechanism for wound-healing than PWD without this particular complication. If the hypothesis is proven correct, this will empower patients and physicians with the diagnostic tests to make early interventions towards avoiding the complications of diabetes.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of diabetes
* Barbadian national
* self reported ethnicity of Black/African descent
* clear knowledge of ulcer history

Exclusion Criteria:

* no clinical diagnosis of diabetes
* non-national of Barbados
* self reported ethnicity not Black/African Descent
* unclear knowledge of ulcer history

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Black Barbadians who are clinically diagnosed as type II diabetes mellitus patients
Sampling Method: Non-Probability Sample
Enrollment: 605 (Estimated)
Dates: Start 2009-12; Primary Completion 2011-06 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Genetic Phenotyping (Haptoglobin and TRAPS) | 18 months

SECONDARY OUTCOMES:
Reactive Hyperemia Index and Augmentation Index | 18 months
Depression | 18 months
Quality of Life | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Robert C Landis, PhD, Principal Investigator — University of the West Indies; Anselm J Hennis, PhD, Study Chair — Univesity of the West Indies; Ian R Hambleton, PhD, Study Chair — University on the West Indies; Andre R Greenidge, BSc, Study Director — University of the West Indies
Locations (1):
- Chronic Disease Research Centre, Bridgetown, Saint Michael, Barbados

REFERENCES:
- [Background] Hennis AJ, Fraser HS, Jonnalagadda R, Fuller J, Chaturvedi N. Explanations for the high risk of diabetes-related amputation in a Caribbean population of black african descent and potential for prevention. Diabetes Care. 2004 Nov;27(11):2636-41. doi: 10.2337/diacare.27.11.2636. PMID 15504998
- [Background] Hambleton IR, Jonnalagadda R, Davis CR, Fraser HS, Chaturvedi N, Hennis AJ. All-cause mortality after diabetes-related amputation in Barbados: a prospective case-control study. Diabetes Care. 2009 Feb;32(2):306-7. doi: 10.2337/dc08-1504. Epub 2008 Nov 4. PMID 18984775